CLINICAL TRIAL: NCT05888142
Title: Exploring the Role of Immersive Virtual Reality in Managing Upper-limb Complex Regional Pain Syndrome in Adults
Brief Title: Using Immersive Virtual Reality to Treat Complex Regional Pain Syndrome in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Mayday Fund (Other)
Responsible Party: Principal Investigator, Miles Fontenot, Resident: School of Medicine: Anesthesiology & Pain Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00015202
Record Dates: First submitted 2023-04-21; First posted 2023-06-05 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Pain, Chronic
Keywords: chronic pain, complex regional pain syndrome, virtual reality, home based, mindfulness, pain neuroscience education
MeSH Terms: conditions — Chronic Pain; Complex Regional Pain Syndromes

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups (exploratory). One group will receive VR more often than the other group. Primary Hypothesis. As planned apriori, collapsing across groups, using a within subject repeated measures ANOVA (or non-parametric equivalent), we predict that compared to pre-treatment, our sample of CRPS (chronic pain) patients will report a significant improvement in the amount of CRPS pain (e.g., less pain) and improved (increased) physical ability/functionality after four months of home-based VR therapy homeworks (four months after baseline) and that they would continue to report significant improvements on an ad-hoc one year post-treatment followup. Secondary hypothesis. CRPS patients would show reduced CRPS hypersensitivity to brief thermal (e.g., cold) stimuli. and reduced CRPS-related co-morbid psychological symptoms after 4 months of home-based VR therapy, and on long term improvements on ad-hoc followup measures one year post-treatment.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants will not be told there is more than one treatment group, but during the consenting process each participant will be fully informed about the treatment they will personally receive. The statistician will not be told which group received more treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Roosevelt "in clinic VR" (Active Comparator): During the "in clinic" training phase of the study, patients in this group will receive VR physical therapy exercises "in clinic" only (no homeworks during training). After the training phase, all patients will do VR homeworks, including VR exercises and VR mindfulness.
  Interventions: Behavioral: in clinic pain VR reduction exercises
- Roosevelt "in Clinic VR" + "VR homeworks" (Experimental): During the training phase, patients in this group will receive VR physical therapy exercises "in clinic". In addition, during the training phase, they will also take a VR system home and will be encouraged to do VR homeworks at home. After the training phase, all patients will do VR homeworks, including VR exercises and VR mindfulness.
  Interventions: Behavioral: In clinic VRpain reduction exercises + VR homeworks

INTERVENTIONS:
Behavioral: in clinic pain VR reduction exercises — During the in clinic training phase, participants will use commercially available VR during "in clinic" VR physical therapy exercises, to help reduce their pain and improve functionality. But this group will not take a VR system home until after completing the in clinic training phase.
  Arms: Roosevelt "in clinic VR"
Behavioral: In clinic VRpain reduction exercises + VR homeworks — During the training phase, participants will use commercially available VR during "in clinic" physical therapy exercises, and during the training phase, they will also receive a VR system they take home and will begin VR homeworks during the traininng phase, to help reduce their pain and improve functionality.
  Arms: Roosevelt "in Clinic VR" + "VR homeworks"

SUMMARY:
This study is designed to test if the use of virtual reality (VR) can improve chronic pain related to CRPS. One way is to use virtual reality. Virtual reality involves looking into a set of goggles and interacting with a computer-simulated world. The use of VR has been shown to be an effective treatment for other pain conditions (Hoffman et al., 2019) and is inexpensive and noninvasive.

DETAILED DESCRIPTION:
Participants will "go into" simple fun pain distracting virtual reality worlds (no previous video game experience needed) that encourages physical movement of the injured limb (e.g., their injured hand). They will also learn some simple daily 10 minute stress reduction, mood lifting mindfulness skills in VR and will receive audio instructions to focus their attention on the sights and sounds, and controlled breathing (Flores et al., 2019).

ELIGIBILITY:
Inclusion Criteria

* adults (18+)
* confirmed diagnosis of either CRPS I or CRPS II of one or both upper limbs (as defined by the Budapest Criteria)
* average pain score in the affected CRPS limb(s) greater than or equal to 3 out of 10
* on a stable treatment plan for 4 weeks prior to the VR intervention phase
* ability to wear a VR head-mounted display
* ability to speak and read English
* ability to provide informed consent.

Exclusion Criteria:

* personal history of severe motion sickness
* severe systemic disease that is a constant threat to life (ASA class IV+)
* prisoners.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2024-08-03 (Actual); Study Completion 2024-08-03 (Actual)

PRIMARY OUTCOMES:
The Patient Global Impression of Change scale (PGIC), regarding CRPS pain. | Change from baseline to 16 weeks
  This self-report measure. reflects a patient's belief about the efficacy of treatment.
  Compared with before receiving VR therapy, how would you describe your pain related to CRPS now overall? 7 point scale from - 3 to + 3 (-3 = very much worst, +3 = very much better). This is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change in CRPS pain as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
The Patient Global Impression of Change scale (PGIC), regarding CRPS pain. | Change from baseline to 1 year post-treatment
  This self-report measure. reflects a patient's belief about the efficacy of treatment.
  Compared with before receiving VR therapy, how would you describe your pain related to CRPS now overall? 7 point scale from - 3 to + 3 (-3 = very much worst, +3 = very much better). This is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change in CRPS pain as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
The Patient Global Impression of Change scale (PGIC), regarding functionality/physical abilities. | Change from baseline to 16 weeks
  This self-report measure reflects a patient's belief about the efficacy of treatment.
  Compared with before receiving VR therapy, how would you describe your physical abilities now overall? 7 point scale from - 3 to + 3 (-3 = very much worst, +3 = very much better). This is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change in physical abilities as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
The Patient Global Impression of Change scale (PGIC), regarding functionality/physical abilities. | Change from baseline to one year post-treatment
  This self-report measure reflects a patient's belief about the efficacy of treatment.
  Compared with before receiving VR therapy, how would you describe your physical abilities now overall? 7 point scale from - 3 to + 3 (-3 = very much worst, +3 = very much better). This is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change in physical abilities as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."

SECONDARY OUTCOMES:
The Central Sensitization Inventory (CSI). | Change from baseline to 16 weeks
  The Central Sensitization Inventory (CSI) is a self-report screening instrument designed to measure exaggerated pain sensitivity. 25 questions, patients answer "never, rarely sometimes, often, always".
The Central Sensitization Inventory (CSI). | Change from baseline to one year post-treatment
  The Central Sensitization Inventory (CSI) is a self-report screening instrument designed to measure exaggerated pain sensitivity. 25 questions, patients answer "never, rarely sometimes, often, always".
CES-D Center for Epidemiologic Studies Depression Scale (CES-D), NIMH. | Change from baseline to 16 weeks
  20 self-rating questions about how depressed the patient has felt during the past week: rarely, a little of the time, a moderate amount of time, most or all of the time.
CES-D Center for Epidemiologic Studies Depression Scale (CES-D), NIMH. | Change from baseline to one year post-treatment
  20 self-rating questions about how depressed the patient has felt during the past week: rarely, a little of the time, a moderate amount of time, most or all of the time.
Mindfulness. | Change from baseline to 16 weeks.
  Mindfulness. Using a single item graphic rating scale, Patients are asked "how mindful were you during the past week? (on a zero to 10 scale where 0 is not mindful at all, and 10 = completely present in the moment, 100% of the time).
Mindfulness. | Change from baseline to one year post-treatment
  Mindfulness. Using a single item graphic rating scale, Patients are asked "how mindful were you during the past week? (on a zero to 10 scale where 0 is not mindful at all, and 10 = completely present in the moment, 100% of the time).
Pain Catastrophizing Scale. | Change from baseline to 16 weeks.
  Pain Catastrophizing Scale. Patients answer 13 questions about thoughts and feelings they have when they are in pain. Not at all, to a slight degree, to a moderate degree, to a great degree, all the time.
Pain Catastrophizing Scale. | Change from baseline to one year post-treatment
  Pain Catastrophizing Scale. Patients answer 13 questions about thoughts and feelings they have when they are in pain. Not at all, to a slight degree, to a moderate degree, to a great degree, all the time.
The 8-item PROMIS Sleep Disturbance Short Form. | Change from baseline to 16 weeks.
  The 8-item PROMIS Sleep Disturbance Short Form assesses the sleep quality in the past 7 days, in individuals age 18 and older. Patients rate each question as Very poor, poor, fair, good, very good.
The 8-item PROMIS Sleep Disturbance Short Form. | Change from baseline to one year post-treatment.
  The 8-item PROMIS Sleep Disturbance Short Form assesses the sleep quality in the past 7 days, in individuals age 18 and older. Patients rate each question as Very poor, poor, fair, good, very good.
Quickdash (measure of physical function). | Change from baseline to 16 weeks
  Patients rate their ability to do a number of activities, 11 questions. QuickDASH uses 11 items to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb.
Quickdash (measure of physical function). | Change from baseline to one year post-treatment.
  Patients rate their ability to do a number of activities, 11 questions. QuickDASH uses 11 items to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb.
Tampa Scale for Kinesiophobia. | Change from baseline to 16 weeks.
  Patients answer 17 questions about their fear of movement by responding "strongly disagree, disagree, agree, or strongly agree".
Tampa Scale for Kinesiophobia. | Change from baseline to one year post-treatment.
  Patients answer 17 questions about their fear of movement by responding "strongly disagree, disagree, agree, or strongly agree".

CONTACTS AND LOCATIONS:
Overall Officials: Miles Fontenot, MD, Ph.D, Principal Investigator — University of Washington
Locations (1):
- University of Washington (only CRPS patients are eligible), Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
we will analyze and publish our results.

REFERENCES:
- [Background] Hoffman HG, Patterson DR, Rodriguez RA, Pena R, Beck W, Meyer WJ. Virtual Reality Analgesia for Children With Large Severe Burn Wounds During Burn Wound Debridement. Front Virtual Real. 2020 Dec;1:602299. doi: 10.3389/frvir.2020.602299. Epub 2020 Dec 10. PMID 33585833
- [Background] Flores A, Linehan MM, Todd SR, Hoffman HG. The Use of Virtual Reality to Facilitate Mindfulness Skills Training in Dialectical Behavioral Therapy for Spinal Cord Injury: A Case Study. Front Psychol. 2018 Apr 23;9:531. doi: 10.3389/fpsyg.2018.00531. eCollection 2018. PMID 29740365
- [Background] Ferguson L, Scheman J, Patient global impression of change scores within the context of a chronic pain rehabilitation program, The Journal of Pain, Volume 10, 2009, S73. ISSN 1526-5900, https://doi.org/10.1016/j.jpain.2009.01.258.
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Background] Neblett R, Cohen H, Choi Y, Hartzell MM, Williams M, Mayer TG, Gatchel RJ. The Central Sensitization Inventory (CSI): establishing clinically significant values for identifying central sensitivity syndromes in an outpatient chronic pain sample. J Pain. 2013 May;14(5):438-45. doi: 10.1016/j.jpain.2012.11.012. Epub 2013 Mar 13. PMID 23490634
- [Background] Radloff, L. S. (1977). The CES-D scale: A self report depression scale for research in the general population. Applied Psychological Measurements, 1, 385-401.
- [Background] Sullivan, M. J. L., Bishop, S. C., and Pivik, J. (1995). The Pain Catastrophizing Scale: Development and validation. Psychol Assess. 7: 524-532.
- [Background] Yu L, Buysse DJ, Germain A, Moul DE, Stover A, Dodds NE, Johnston KL, Pilkonis PA. Development of short forms from the PROMIS sleep disturbance and Sleep-Related Impairment item banks. Behav Sleep Med. 2011 Dec 28;10(1):6-24. doi: 10.1080/15402002.2012.636266. PMID 22250775
- [Background] Beaton DE, Wright JG, Katz JN; Upper Extremity Collaborative Group. Development of the QuickDASH: comparison of three item-reduction approaches. J Bone Joint Surg Am. 2005 May;87(5):1038-46. doi: 10.2106/JBJS.D.02060. PMID 15866967
- [Background] Vlaeyen JW, Kole-Snijders AM, Rotteveel AM, Ruesink R, Heuts PH. The role of fear of movement/(re)injury in pain disability. J Occup Rehabil. 1995 Dec;5(4):235-52. doi: 10.1007/BF02109988. PMID 24234727
- [Derived] Fontenot MR, Curatolo M, Stacey BR, Flor H, Hoffman HG. Sustained symptom reduction in complex regional pain syndrome with a novel home-based virtual reality program: a pilot study. Front Neurol. 2025 Dec 8;16:1622897. doi: 10.3389/fneur.2025.1622897. eCollection 2025. PMID 41438885